CLINICAL TRIAL: NCT04965805
Title: The Treatment of Chronic Wounds With the Cold Plasma Jet kINPen® Med Versus Best Practice Wound Dressings: a Multicenter, 2-Armed, Randomized, Open-label, Prospective, Non-inferiority Clinical Trial
Brief Title: Cold Plasma Jet kINPen Med Versus Best Practice Wound Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University Teaching Hospital, Feldkirch, Austria (Other)
Collaborators: neoplas Med (Unknown)
Responsible Party: Principal Investigator, Robert Strohal, Primarius Professor Dr., Federal University Teaching Hospital, Feldkirch, Austria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6/6-2-19
Record Dates: First submitted 2021-07-05; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Wounds
Keywords: Plasma; Dressings
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study is a double-center, two-armed, randomized, prospective, non-inferiority, clinical comparative trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold plasma jet (Experimental): The treatment scheme of the cold plasma jet will be applied in the following manner, quantity and frequency: Cold plasma is always applicated for 30 seconds/ cm^2 wound size. Wounds will be treated three times in the first week, twice in the second week and once per week in the following observation period. In case of locally infected ulcers, treatment will be performed 1x per day during the first week and afterwards in the same manner as in non-infected ulcers. After application of cold plasma, the wound will be covered with Adaptic perforated gauze and a non-active dressing.
  Interventions: Device: cold plasmaJet kINPen Med
- Best Practice wound dressings (Active Comparator): Immediately after dressing removal, the wound will be cleaned with a physiological saline solution soaked swab. In case of locally infected wounds, an antiseptic will be used instead of the physiological saline solution. Subsequently, a wound phase-adapted primary dressing will be applied according to the experience of the practitioner and, if necessary, the wound will be covered with a secondary dressing according to the experience of the practitioner as well. In case of locally infected wounds, silver dressings can be applied. The dressing will be changed at least every 2nd day and on weekends every 3rd day; in case of locally infected wounds, dressings will be changed daily. Dressing changes beyond visits can also be performed by the general practitioner, a nursing service, or by the participant him- or herself.
  Interventions: Device: Best practice wound dressings

INTERVENTIONS:
Device: cold plasmaJet kINPen Med — experimental, non-inferiority
  Arms: Cold plasma jet
Device: Best practice wound dressings — comparative,
  Arms: Best Practice wound dressings

SUMMARY:
Within the treatment of chronic wounds the main objective is to analyze the wound healing properties with cold plasma (cold plasma jet kINPen® Med) compared to wound phase-adapted best practice wound dressings. Especially, close attention is paid to the development of the different phases of the chronic wounds until healing during the study.

DETAILED DESCRIPTION:
Cold plasma jet arm: Immediately after removal of the dressing, the wound will be cleaned with a physiological saline solution soaked swab. If > 30% fibrin coating or dry necrosis remaines after cleaning, debridement is required before treatment. The treatment scheme of the cold plasma jet will be applied in the following manner, quantity and frequency: Cold plasma is always applicated for 30 seconds/ cm^2 wound size. Wounds will be treated three times in the first week, twice in the second week and once per week in the following observation period. In case of locally infected ulcers, treatment will be performed 1x per day during the first week and afterwards in the same manner as in non-infected ulcers. After application of cold plasma, the wound will be covered with Adaptic perforated gauze and a non-active dressing. Dressing change will be performed after treatment and at least every 2nd day, on weekends every 3rd day; in the case of locally infected wounds, dressings will be changed daily. The application of cold plasma will be performed always by the examiner. Dressing changes beyond visits can also be performed by the general practitioner, a nursing service or by the participant him- or herself.

Best Practice treatment arm: Immediately after dressing removal, the wound will be cleaned with a physiological saline solution soaked swab. In case of locally infected wounds, an antiseptic will be used instead of the physiological saline solution. Subsequently, a wound phase-adapted primary dressing will be applied according to the experience of the practitioner and, if necessary, the wound will be covered with a secondary dressing according to the experience of the practitioner as well. In case of locally infected wounds, silver dressings can be applied. The dressing will be changed at least every 2nd day and on weekends every 3rd day; in case of locally infected wounds, dressings will be changed daily. Dressing changes beyond visits can also be performed by the general practitioner, a nursing service, or by the participant him- or herself.

In case of a venous leg ulcer, a modern compression system will be applied for compression in both study arms.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study, participants must meet the following criteria:

  * chronic wounds of any origin or wound phase, including locally infected chronic ulcers
  * wound size up to 20x10 cm
  * wounds without visible tendon or bone
  * participant age between 18 95 years

Exclusion Criteria:

* • acute wounds

  * in case of multiple wounds, only one wound will be assigned as study wound
  * wounds with > 30 percentage necrotic eschar
  * pregnant or breastfeeding women or women of childbearing age
  * participants with intake of antibiotics within one week before the start of the enrollment
  * allergy or intolerance against a primary or secondary dressing
  * allergy or intolerance against cold plasma
  * participation in any other clinical trial up to one month prior to study enrollment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Percentage of the Sum of Granulation Tissue on the Wound | Day 42 ±2
  At baseline (Day 0) and each subsequent visit, the total amount of granulation tissue of each wound will be documented as percentage of wound area. The entire circumference of the ulcer will be traced, then divided into four equal parts (one quadrant corresponding to 25 percentage), and the amount of granulation tissue will be measured using a ruler. The percentage corresponding to the amount will be determined mathematically.

SECONDARY OUTCOMES:
Wound size reduction and healing | Day 42 ±2
  The dynamic of the wound size in cm^2 is measured by a digital automated system.

OTHER OUTCOMES:
Change Infection PGA Score | Day 0 to Day 42 ±2
  At baseline (Day 0) and each subsequent visit, clinical signs of a local infection will be documented according to the Physician Global Assessment (PGA) Score:
  infection PGA 4: very strong infection PGA 3: strong infection PGA 2: moderate infection PGA 1: mild infection PGA 0: absent
Change ph of the wound | Day 3 to Day 42 ± 2
  Prior to each dressing change, the pH value of the wound bed or the central wound fluid will be measured with an adjusted pH meter calibrated to pH 7.
Change Exudate level | Day 3 to Day 42 ± 2
  The amount of wound exudate will be determined by the study practitioner and quantified on a scale from 0 to 4 at the below specified study visits:
  4: highly exudative 3: strong 2: moderate
  1: mild 0: absent
Participant's Sensation of the Application of the Cold Plasma Jet | Day 3
  In the cold plasma jet arm, the participants will be asked to rate their sensation after the cold plasma treatment on a scale from 1 to 4:
  4 - very unpleasant (severe pain, burning sensation) 3 - uncomfortable 2 - no specific sensibility
  1 - pleasant feeling (e.g. cooling)
Local tolerability | Day 35 ± 2
  During each dressing change after Day 0, the tolerability of the treatment substances used will be evaluated according to the following parameters:
  * no problem (e. g., no maceration, wound deterioration or blisters)
  * emergence or exacerbation of
    * erythema
    * maceration
    * blisters
    * congestion of exudate

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Academic Teaching Hospital Feldkirch, Feldkirch, Vorarlberg, Austria

IPD SHARING:
Plan to Share IPD: No